CLINICAL TRIAL: NCT06279442
Title: Adrenal Project: Clinical and Epidemiological Characterization of Adrenocortical Carcinoma in a Brazilian Cohort
Status: Recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0723
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma Adrenal; Carcinoma, Adrenocortical Recurrent
Keywords: Carcinoma adrenocortical
MeSH Terms: conditions — Adrenal Cortex Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective observational cohort study. The clinical, pathological and treatment data of participants identified with adrenocortical carcinoma from the year 2000 onwards will be evaluated. Participants recruited for this study will be identified at the participating sites.

DETAILED DESCRIPTION:
Adrenocortical carcinoma is one of the rarest neoplasms in the world. In Brazil, especially in the South and Southeast regions, the incidence of adrenocortical tumors is around 15 times higher than in the rest of the world, largely attributed to the significant prevalence of the TP53-R337H germline mutation in this population. In view of this characteristic, the clinical and epidemiological characterization of this cohort, as well as the identification of prognostic factors, is of great importance. The starting point for this project was the cohort of 66 participants with adrenal carcinoma included in the final project of the medical residency in clinical oncology at the A.C. Camargo Cancer Center by student Rafael Haikal dos Santos Abduch. The aim is to include case studies from the main Brazilian site that have followed up and treated patients with adrenal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old;
* Diagnosis of adrenocortical carcinoma with at least one clinical evaluation at the reference institution;
* Initial diagnosis or recurrence from the year 2000 onwards.

Exclusion Criteria:

* Participants with insufficient clinical or pathological data in the medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be included from 150 participants diagnosed with adrenocortical carcinoma who meet the study's inclusion and exclusion criteria. Data will be collected from the medical records of the included research sites throughout Brazil.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Demographic Characterization of Adrenocortical Carcinoma in Brazil | Throughout the study period, an average of 18 months.
  This measure aims to capture essential demographic attributes of individuals in Brazil diagnosed with adrenocortical carcinoma. It will include details such as age distribution in years, gender representation, geographic distribution, height in meters, weight in kilograms, as well as racial and ethnic demographics . These insights will contribute to a comprehensive understanding of the demographic landscape of adrenocortical carcinoma within the Brazilian population.
Clinical Characterization of Adrenocortical Carcinoma in Brazil | Throughout the study period, an average of 18 months.
  This measure aims to capture essential clinical attributes of individuals in Brazil diagnosed with adrenocortical carcinoma. It will include relevant clinical factors such as tumor stage, hormone secretion status, and treatment modalities. These insights will contribute to a comprehensive understanding of the clinical landscape of adrenocortical carcinoma within the Brazilian population.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Shizue Tariki, Principal Investigator — Latin American Cooperative Oncology Group
Locations (10):
- Brazil (10):
  - Pronutrir - Suporte Nutricional e Quimioterapia, Fortaleza, Ceará
  - Hospital do Câncer do Maranhão Dr. Tarquínio Lopes Filho, São Luís, Maranhão
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Santa Joana Recife (Instituto Américas PE), Recife, Pernambuco
  - UOPECCAN - Hospital do Câncer de Cascavel, Cascavel, Santa Catarina
  - FUNFARME - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - HAOC - Hospital Alemão Oswaldo Cruz, São Paulo
  - A.C. Camargo Cancer Center, São Paulo